CLINICAL TRIAL: NCT06756659
Title: Comparison of the Effectiveness Between Home-based Cardiac Rehabilitation With Spot-jogging and Outpatient Center-Based Cardiac Rehabilitation in Patients With Heart Failure.
Brief Title: Home-based Cardiac Rehabilitation With Spot-jogging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202406057RIND
Record Dates: First submitted 2024-12-08; First posted 2025-01-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Cardiac Rehabilitation
Keywords: HF; CR
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based cardiac rehabilitation group (Experimental): All participants will undergo spot jogging cardiopulmonary exercise test and six-minute walking test. The home-based spot jogging cardiac rehabilitation group will receive exercise intensity guidance in the outpatient cardiac rehabilitation room for 30 minutes of spot jogging and treadmill exercise during the first, fourth, and seventh weeks, and will perform moderate-intensity spot jogging for 30 minutes twice a week at home.
  Interventions: Other: Home-based spot jogging
- outpatient center-based cardiac rehabilitation group (Active Comparator): All participants will undergo spot jogging cardiopulmonary exercise test and six-minute walking test. The outpatient center-based cardiac rehabilitation group will perform moderate-intensity stationary bike or treadmill exercise for 30 minutes twice a week in the outpatient cardiac rehabilitation room.
  Interventions: Other: Center-based exercise training

INTERVENTIONS:
Other: Center-based exercise training — All participants will undergo a spot jogging cardiopulmonary exercise test and a six-minute walking test. The outpatient center-based cardiac rehabilitation group will perform moderate-intensity stationary biking or treadmill exercise for 30 minutes, twice a week, under the supervision of a physical therapist in the outpatient cardiac rehabilitation room.
  Arms: outpatient center-based cardiac rehabilitation group
Other: Home-based spot jogging — The home-based spot jogging cardiac rehabilitation group will receive exercise intensity guidance in the outpatient cardiac rehabilitation room for 30 minutes of spot jogging and treadmill exercise during the first, fourth, and seventh weeks. They will then perform moderate-intensity spot jogging at home for 30 minutes, twice a week, at a perceived exertion level of 13 out of 20 on the RPE scale.
  Arms: home-based cardiac rehabilitation group

SUMMARY:
The first purpose of this study is to investigate the physiological changes of heart failure patients during cardiopulmonary exercise test with spot jogging and compare them with the standard stationary bike cardiopulmonary exercise test. The second one is to compare the effect between home-based cardiac rehabilitation using different step frequency and toe lift or not to adjust spot jogging intensity and outpatient center-based cardiac rehabilitation for heart failure patients.

DETAILED DESCRIPTION:
This is a pilot, prospective, randomized controlled trial design. We will recruit 40 heart failure patients aged over 18 year-old who have completed stationary bike cardiopulmonary exercise test and was referred to phase II cardiac rehabilitation. After providing informed consent, participants will be randomly assigned to either the home-based cardiac rehabilitation group or the outpatient center-based cardiac rehabilitation group. All participants will undergo spot jogging cardiopulmonary exercise test and six-minute walking test. The home-based spot jogging cardiac rehabilitation group will receive exercise intensity guidance in the outpatient cardiac rehabilitation room for 30 minutes of spot jogging and treadmill exercise during the first, fourth, and seventh weeks, and will perform spot jogging for 30 minutes twice a week at home. The outpatient center-based cardiac rehabilitation group will perform stationary bike or treadmill exercise for 30 minutes twice a week in the outpatient cardiac rehabilitation room. Both groups will achieve their target heart rate or 13 in rating perceived exertion. After 18 exercise sessions, participants will undergo stationary bike exercise test and six-minute walking test again.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients aged over 18 year-old who have completed stationary bike cardiopulmonary exercise test and was referred to phase II cardiac rehabilitation.

Exclusion Criteria:

* Atrial fibrillation
* Other neurological or musculoskeletal issues that affect physical activity.
* Undergoing dialysis.
* Having a pacemaker.
* Unable to cooperate in completing cardiopulmonary exercise testing.
* Do not agree to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test | baseline at enrollment and the end of treatment at 9 weeks (after 18 exercise sessions)

SECONDARY OUTCOMES:
Six-minute walking test | baseline at enrollment and the end of treatment at 9 weeks (after 18 exercise sessions)
36-Item Short Form Health Survey | baseline at enrollment and the end of treatment at 9 weeks (after 18 exercise sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ikenaga M, Yamada Y, Kose Y, Morimura K, Higaki Y, Kiyonaga A, Tanaka H; Nakagawa Study Group. Effects of a 12-week, short-interval, intermittent, low-intensity, slow-jogging program on skeletal muscle, fat infiltration, and fitness in older adults: randomized controlled trial. Eur J Appl Physiol. 2017 Jan;117(1):7-15. doi: 10.1007/s00421-016-3493-9. Epub 2016 Nov 15. PMID 27848017